CLINICAL TRIAL: NCT02603354
Title: Efectiveness of a Brief Protocol by a Low (6%) Concentration Gel Peroxide Hydrogen of Teeth Bleaching
Acronym: Brief6%
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Eduardo Fernandez, Prof. Dr. Eduardo Fernández, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15/001a
Record Dates: First submitted 2015-11-08; First posted 2015-11-11 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Tooth Discoloration
MeSH Terms: conditions — Tooth Discoloration

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 3x12 m peroxide gel tooth bleaching 6% (Active Comparator): bleaching with 6% hydrogen peroxide 3 times of 12 minutes session for in office bleaching teeth
  Interventions: Drug: peroxide gel tooth bleaching 6%
- 1-36 m peroxide gel tooth bleaching 6% (Experimental): bleaching with 6% hydrogen peroxide 1 time of 36 minutes session for in office bleaching teeth
  Interventions: Drug: peroxide gel tooth bleaching 6%

INTERVENTIONS:
Drug: peroxide gel tooth bleaching 6% — gel of hygrogen peroxide for teeth bleaching in a low concentration (6%)
  Other Names: bleaching gel

SUMMARY:
The purpose of this clinical study was to evaluate, the effectiveness and sensitivity post-treatment of a 6% hydrogen peroxide with nitrogen-doped titanium dioxide light activated bleaching agent, the impact of shorter interval times on tooth sensitivity and to compare the efficacy with 2 different application protocols. This is a clinical randomized double-blind split-mouth study. 31 patients were treated with: one upper hemi arcade with one application of 36 minutes and the other hemi arcade with 3 applications of 12 minutes each with a 6% hydrogen peroxide. Two sessions were appointed with 48h of intervals between them. Tooth colour was registered by VITA Classical amd VITA Bleach guide by two blinded assessors in the beginning, immediately after each session. Tooth colour variation and sensitivity were compared between both application protocols

DETAILED DESCRIPTION:
This was a randomized, triple-blinded (patients, evaluator, and statistician), and split-mouth design (one hemiarcade was treated by 2 different protocol applications) following nonprobability sampling. The patients were invited to participate in the study through posters posted around the city or recruited from participants in other studies in the same department, who were contacted by email or phone.

A total of 155 patients were examined in a dental chair to check if they met the inclusion and exclusion criteria. The patients included in this study were over 18 years old and selected with the following inclusion criteria: anterior teeth without restorations, previous bleaching procedures, cervical lesions, or dental pain. Patients who were pregnant or lactating, had moderate or severe fluorosis, tetracycline stains, orthodontic treatment, periodontal disease, orofacial tumors, trauma, or tooth malformation, or were taking analgesic, anti-inflammatory, or antibiotic drugs were excluded.

Two trained operators (restorative dentistry professors) performed the bleaching treatments. A third participant that did not have contact with the patients was responsible for conducting the randomization. The allocation of the hemiarcade in the groups was performed by random drawing using Microsoft Excel 2010 (Microsoft, Redmond, Washington, USA) from coding assigned to each participant. There were two experimental groups: Group A acted as a control, and hydrogen peroxide whitening compound was applied at a concentration of 6% to the upper hemiarcade with a convetional protocol application of 3 times of 12 minutes. Group B was the experimental group, in which the other upper hemiarcade was treated with 6% and a reduce application protocol of 1 times of 36 minutes , the both hemiarcades were bleached with the same compound catalyzed by titanium oxide nanoparticles and activated by blue hybrid light and an infrared laser.

Sample size calculation The primary outcome of this study was the efficacy determined by color alteration (ΔE). Previous studies showed that the use of in-office bleaching agent containing hydrogen peroxide (HP35) with or without LED/Laser light leads to a ΔE value of 7.0-2.0 after two bleaching sessions. In order to have an 80% chance of detecting significance at the level of 5%, and considering an increase in the primary outcome measure from 7 in the control group to 5 in the experimental group, a minimum of 16 participants would be required in each group. Due to a higher dropout rate in the last two clinical studies of our research group, The investigators decided to add 80% more patients, which led to 30 patients in each group.

Bleaching protocol In each session, volunteers received prophylaxis with pumice powder and water. Then, gingival tissue was protected using a light-cured resin gum barrier applied according to the manufacturer's instructions (Lase Protect - DMC, São Carlos, SP, Brazil). The bleaching agent was prepared by mixing hydrogen peroxide and thickening compounds according to the manufacturer's instructions (with 3 peroxide drops for 1 drop of thickener). The resultant gel was distributed uniformly on the upper hemiarcade surfaces of the teeth. A total of 8 teeth between the first premolars were bleached for each patient. In each bleaching session, the bleaching gels were applied three times for 12 minutes each and the other hemiarcade only for a 36 minutes by session. In each application, the surface of the gel was light activated with continuous irradiance using LED/laser light with a total power of 1800 mW (Whitening Lase Plus - DMC Equipamentos, São Carlos, SP, Brazil). Three bleaching sessions were completed for the patients, and the interval between sessions was 2 days.

Efficacy evaluation (E) Objective evaluation Two calibrated evaluators (Kappa=0.85) were used to measure the tooth color for the baseline (T0), immediately after the first (T1), second (T2), and one week (T3) and one month after the last session (T4). The color evaluation was obtained from an area of 6 mm located in the middle third of the labial surface of the left and right central incisors. To standardize this evaluation, an impression of the maxillary arch was taken to make a guide using high-putty silicone (Zetaplus, Zhermack, Badia Polesine, Rovigo, Italy). A window was created on the labial surface in the middle third of the central incisor using a device with well-formed borders and a 3-mm radius corresponding to the reflectance of the spectrophotometer (Vita EasyShade Compact, VITA Zahnfabrik, Bad Säckingen, Germany). The shade was determined using the obtained parameters L*, a*, and b*. The color alteration after each session was given by the differences between the values obtained at the session and the baseline (∆E). ∆E was calculated using the following formula: ΔE = [(ΔL*)2 + (Δa*)2 + (Δb*)2]1/2 .

Subjective evaluation For the subjective evaluation, the 16 tabs of the shade guide (Vita Classic, Vita Zahnfabrik) were arranged from the highest (B1) to the lowest (C4) value. Although this scale is not linear in the truest sense, The investigators treated the changes as continuous with a linear ranking, as was done in several clinical trials of dental bleaching. Two calibrated evaluators (Kappa=0.85) recorded the shade of the upper central left and right incisors at baseline with the same periods as the objective evaluation.

The investigators checked the color in the middle third area of the labial surface of the anterior central incisor according to the American Dental Association guidelines. The investigators calculated the color changes from the beginning of the active phase through the individual recall times by the change in the number of shade guide units (ΔSGU), which occurred toward the lighter end of the value-oriented list of shade tabs. In the event that the operators disagreed on color matching, a consensus was reached prior to dismissing the patient.

Tooth sensitivity evaluation (S) Tooth sensitivity was characterized by the variables occurrence, intensity, and type. These data were obtained by self-completed form and clinical evaluation during the session and immediately by VAS (Visual Analogue Scale). For the VAS, The investigators instructed the participants to place a line perpendicular to a 10-mm-long line with zero at one end indicating ''no TS'' and the other end indicating ''unbearable TS.'' The occurrence was analyzed according to whether sensitivity was reported. The intensity was measured at four levels according to a verbal scale: 1=none, 2=mild, 3=moderate, 4=considerable, and 5=severe. The volunteers were instructed to fill out a form for each bleaching session and for the following days between sessions in case of sensitivity in any of the bleached teeth at any time.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients with Anterior teeth without restorations, previous bleaching procedures, cervical lesions, or dental pain

Exclusion Criteria:

* Pregnant or lactating,
* Had moderate or severe fluorosis,
* Tetracycline stains,
* Orthodontic treatment,
* Periodontal disease,
* Orofacial tumors,
* Trauma,
* Tooth malformation,
* Were taking analgesic, anti-inflammatory, or antibiotic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-03; Primary Completion 2015-04 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Efectiveness by color difference ( using the spectrophotometer Vita Easy Shade) | 1 month
  The shade was determined using the obtained parameters L*, a*, and b* by Spectrophotometer . The color alteration after each session was given by the differences between the values obtained at the session and the baseline (∆E). ∆E was calculated using the following formula: ΔE = [(ΔL*)2 + (Δa*)2 + (Δb*)2]1/2 .

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Fernandez, PhD, Study Director — University of Chile
Locations (1):
- Eduardo Fernandez, Santiago, N/A = Not Applicable, Chile

REFERENCES:
- [Background] Martin J, Vildosola P, Bersezio C, Herrera A, Bortolatto J, Saad JR, Oliveira OB Jr, Fernandez E. Effectiveness of 6% hydrogen peroxide concentration for tooth bleaching-A double-blind, randomized clinical trial. J Dent. 2015 Aug;43(8):965-72. doi: 10.1016/j.jdent.2015.05.011. Epub 2015 Jun 6. PMID 26057085